CLINICAL TRIAL: NCT04997603
Title: Sleep, Physical Activity, and Dietary Habits Among High School Student-athletes and Non-athletes During an Academic Semester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1914
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sleep Quantity; Sleep Efficiency
Keywords: sleep; adolescent; Fitbit; accelerometer; athlete; stress; students

STUDY DESIGN:
Intervention Model Description: Fitbit accelerometers are distributed to both groups, student athletes and non-athletes who continue to live their lives as usual during the 2 week monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Athletes wearing an accelerometer continuously for 2 weeks (Other): High school students: 50% male, 50% female
  Interventions: Other: Accelerometer
- Non-athletes wearing an accelerometer continuously for 2 weeks (Other): High school students: 50% male, 50% female
  Interventions: Other: Accelerometer

INTERVENTIONS:
Other: Accelerometer — Fitbit brand

SUMMARY:
Adolescent's poor sleep habits have been linked to adverse outcomes. Recent advances in activity tracking have provided researchers with cost-effective and non-invasive measurements of sleep in a free-living environment. The primary objective is to determine the mean differences in Fitbit accelerometer sleep quantity (mins) between High School student-athletes and non-athletes during a competitive academic semester over continuous monitoring for two weeks.

DETAILED DESCRIPTION:
Secondary objectives are to measure and determine:

* If a relationship exist between self-reported Pittsburgh Sleep Quality Index (PSQI) sleep scores and Perceived Stress Scale (PSS) scores compared to mean Fitbit accelerometer sleep quantity and efficiency (sleep quality) based on heart rate, time awake or restless over two weeks
* If dietary habits have a significantly correlated relationship to subject group, sleep quantity, sleep efficiency and steps/day
* If mean differences exist in Fitbit steps counted between student-athletes and non-athletes over two weeks
* If a relationship exists between mean Fitbit accelerometer steps counted and mean sleep quantity and efficiency over two weeks

All Fitbits are monitored remotely by the Principal investigator. This is a fully remote study (no physical study sites). Participants are recruited from 3 high schools (IRB approved). Consent, study forms and other e-mail communication and texting is directly between the participant and the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. High-school student-athletes and non-athletes ages 15-18 y
2. Enrolled in at least 6 academic credit hours from the same high school
3. Willing and able to wear wrist-worn Fitbit continuously for 14 days
4. Parental consent will be needed for minors (<18 years old)
5. Student-athletes need to be competing in a high school recognized sport during the study period

Exclusion Criteria:

1. Individual has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with the project/study protocol, which might confound the interpretation of the project/study results or put the person at undue risk
2. Those with a medical history that would interfere with the results of this study.
3. Under the care of a physician
4. Skin sensitivities
5. Sleep disorders
6. Using prescription medications that would impact sleep
7. Pregnant
8. Smoker
9. Drug or alcohol user
10. Not able to wear wrist-worn Fitbit continuously for 14 days
11. Non-athletes must not be in an organized sport
12. Lack of proficiency in English
13. Lack of proficiency or access to the internet and email address
14. Are not employed by, or have a parent, guardian or other immediate family member employed by, a company that manufactures any products that compete with any Gatorade products. If you are unsure if a company would be considered a competitor to Gatorade, please let the study investigator know the name of the other company and the nature of your relationship to that company before you sign this form
15. No participation in another clinical trial within the past 30 days, and no participation in a PepsiCo protocol within the past 6 months.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Fitbit mean sleep quantity | Worn for two continuous weeks
  Measured in minutes. More minutes are better.
Fitbit mean sleep efficiency | Worn for two continuous weeks
  Measured as a percentage (0-100% score representing sleep quality based on heart rate, time awake or restless, and sleep stages). Higher percentage is better.

SECONDARY OUTCOMES:
Fitbit steps counted | Two weeks of continuous Fitbit monitoring
  Physical activity measure. More steps are better.
Subjective sleep (PSQI) scores | Two weeks of continuous Fitbit monitoring
  Subjective sleep PSQI (Pittsburgh Sleep Quality Index) scores (0-21). Higher scores are worse.
Subjective stress (PSS) scores | Two weeks of continuous Fitbit monitoring
  Perceived stress PSS (Perceived Stress Scale) scores (0-40). Higher scores are worse.
Dietary REAP | Two weeks of continuous Fitbit monitoring
  Rapid Eating Assessment for Patients (REAP) scores (30-89). Higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Corey T Ungaro, Principal Investigator — PepsiCo Global R&D, Gatorade Sports Science Institute (GSSI)
Locations (4):
- United States (4):
  - Gatorade Sports Science Institute (GSSI), Barrington, Illinois
  - Belton High School, Belton, Texas
  - McGregor High School, McGregor, Texas
  - Lake Belton High School, Temple, Texas

IPD SHARING:
Plan to Share IPD: No